CLINICAL TRIAL: NCT02057445
Title: A Multicenter Pilot Study of Third Party LMP1/2-Specific Cytotoxic T Lymphocytes for Treatment of Patients With Refractory /Relapsed EBV-Associated Lymphoma A Childhood, Adolescent and Young Adult Lymphoma Cell Therapy Consortium (LCTC) Multicenter Clinical Trial
Brief Title: 3rd Party LMP1/2-Specific Cytotoxic T Lymphocytes for EBV-Associated Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: Children's National Research Institute (Other); Baylor College of Medicine (Other); M.D. Anderson Cancer Center (Other); University of Michigan (Other); University of Utah (Other); City of Hope Medical Center (Other); Ohio University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Principal Investigator, New York Medical College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC-561
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Non-Hodgkins Lymphoma; Hodgkins Lymphoma; Lymphoproliferative Disorder
Keywords: cellular therapy; lymphoma; lymphoproliferative disorder
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoproliferative Disorders; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recipient (Experimental): EBV+ patients will receive 3rd party LMP-CTLs for treatment of EBV infection and/or disease
  Interventions: Drug: EBV CTL's
- Donor (Other): Healthy donors who are EBV+ will be asked to donate 60-120 ml of peripheral blood for development of cell lines to be stored for cell line bank.
  Interventions: Other: Peripheral Blood Donor

INTERVENTIONS:
Drug: EBV CTL's — Eligible patients with a matched cell line will be infused with 3rd party CTLs and monitored for adverse events and response. Patients who show a response and tolerate the infusion well may receive up to 5 infusions total 4-6 weeks apart.
  Arms: Recipient
Other: Peripheral Blood Donor — Donors who are EBV+ and meet the eligibility criteria will be consented to provide 60-120 ml peripheral blood once for future use for this and other clinical trials using 3rd party CTLs.
  Arms: Donor

SUMMARY:
The administration of allogeneic third party derived LMP specific-CTLs (special peripheral blood cells from another person) that are made specific to fight EBV infection) in Children, Adolescents and Young Adults (CAYA) with EBV-associated refractory or relapsed lymphoma will be feasible ( able to be done), safe and well tolerated (no unexpected serious events will occur). In addition, potential donors who are EBV positive will be enrolled to donate peripheral blood to help build a bank of these specific EBV fighting cell lines.

ELIGIBILITY:
Inclusion Criteria:

Patient must be at least 1 year of age.

Patient or the patient's legally authorized guardian must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects), and must sign an informed consent in accordance with the institutional policies approved by the U.S. Department of Health and Human Services.

Patients should have been off other investigational therapy for one month prior to entry in this study.

Patient must have adequate organ function as below:

Adequate renal function defined as:

* Serum creatinine <2.0 x normal, or
* Creatinine clearance or radioisotope GFR > 40 ml/min/m2 or >60 ml/min/1.73 m2 or an equivalent GFR as determined by the institutional normal range

Adequate liver function defined as:

* Total bilirubin <2.0 x normal; and
* SGOT (AST) or SGPT (ALT) <5.0 x normal

Adequate pulmonary function defined as:

- Pulse oximetry >94% in room air. Lansky (< 16yr) or Karnofsky (> 16 yrs) performance status ≥ 50% Life expenctancy ≥ 6 weeks. Women of child bearing age require a negative urine pregnancy test. Clinical status at enrollment to allow tapering of steroids to less than 0.5mg/kg/day prednisone at time of treatment.

4.5 Disease Status (Eligibility) 4.5.1 Any patient, with one or more of the following EBV-positive type II latency or associated disorders, regardless of the histological subtype: Hodgkin lymphoma Non-Hodgkin lymphoma Lymphoproliferative disorder Severe chronic active EBV infection syndrome (SCAEBV), defined as high EBV viral load in plasma or PBMC (> 4000 genomes per μg PBMC DNA) and/or biopsy tissue positive for EBV

The disease needs to be in one of the following stages:

At diagnosis who would be unable to receive conventional chemotherapy or in first relapse AND the patient is not a candidate for HSCT Partial response after conventional therapy. Refractory to conventional therapy for his/her condition. In second or subsequent relapse. Residual disease after autologous, syngeneic or allogeneic HSCT.

All patients entered into the study ideally will have tumor tissue from the original diagnostic specimen and/or relapse reviewed centrally for confirmation of EBV positive disease. If no specimen is available, local pathology report documenting EBV positivity is acceptable. Appropriate immunophenotyping to confirm the diagnosis will be performed. In addition, in situ hybridization for EBV (LMP1, and/or EBER positivity) will be performed. All central morphologic analysis and immunohistochemical/insitu hybridization staining will be performed in the laboratory of Sherrie Perkins and Rodney Miles at the University of Utah.

Donor Eligibility for LMP-CTL Third Party Banking (Aim 2.1.2)

* Donor must be HIV negative.
* Donors must have adequate hematopoietic function defined as absolute neutrophil count > 1000/mm3, hemoglobin > 10 g/dl, and platelet count >50,000/mm3 and be EBV IgG seropositive.
* Donors will have peripheral blood collected for LMP specific CTL production. A minimum of 60 cc of peripheral blood x 2 for a total maximum amount of blood of 120cc, will be collected from the donor (subjects must be at least 12 kg or 24 pounds). (See Appendix B) For donors <18 years a maximum of 3cc/kg blood will be taken in an 8 week period.
* For donors that are to undergo stem cell collection, the peripheral blood for LMP specific CTL production will be collected prior to the stem cell collection and without a specific day specification.
* Donor eligibility must meet criteria as per 21 CFR 1271.

Exclusion Criteria:

Currently receiving any investigational agents or have received any tumor vaccines within previous 4 weeks.

Active acute grade III-IV graft-versus-host disease. Severe refractory intercurrent infection other than EBV. Received alemtuzumab or other anti-Tcell antibody within 28 days. HIV seropositivity. Pregnancy (due to unknown effects of this therapy on a fetus) or lactation. Patients with PTLD post solid organ transplantation eligible for the COG PTLD LMP/CTL protocol.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To determine the safety of giving 3rd party EBV-CTLs | 1 year
  Patients will be monitored for any unexpected adverse events related to investigational product.
To develop a third party bank of LMP-specific CTL | on going
  EBV positive donors will be asked to provide an extra sample of peripheral blood to build a donor bank of EBV-CTLs for this protocol and future use.

SECONDARY OUTCOMES:
To measure the response rate | 1 year
  patients will be followed a year following administration of cells for disease response.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD, Principal Investigator — New York Medical College; Catherine Bollard, MD, Principal Investigator — Children's National Research Institute
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - New York Medical College, Valhalla, New York